CLINICAL TRIAL: NCT00411840
Title: Transplantation of Autologous Mononuclear Bone Marrow Stem Cells in Patients With Peripheral Arterial Disease (TAM-PAD Study)
Brief Title: Novel Therapy of PAD by Combined Transplantation of BMCs
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAM-PAD
Record Dates: First submitted 2006-12-13; First posted 2006-12-15 (Estimated); Last update posted 2006-12-15 (Estimated); Status verified 2006-12

CONDITIONS: Peripheral Arterial Disease
Keywords: stem cell therapy; peripheral arterial disease; limb ischemia
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Infusions, Intra-Arterial

INTERVENTIONS:
Procedure: intraarterial and intramuscular injection of BMCs

SUMMARY:
We analyze the effects of combined intramuscular and intraarterial transplantation of BMCs in patients with PAD. BMCs were transplanted into the ischemic limb.

After 2 and 13 months walking distance and perfusion indices were monitored.

ELIGIBILITY:
Inclusion Criteria:

* severe limb ischemia

Exclusion Criteria:

* infectious disease
* cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2004-07

PRIMARY OUTCOMES:
ABI, walking distance, capillary-venous oxygen saturation, venous occlusion plethysmography

SECONDARY OUTCOMES:
feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Bodo E Strauer, MD, Study Director — Heinrich-Heine University, Duesseldorf
Locations (1):
- Heinrich-Heine-University, Düsseldorf, Germany